CLINICAL TRIAL: NCT00875420
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Phase 2, Multi-Center, Dose-Finding Study to Evaluate the Effects of RAD1901 in the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: A Study to Evaluate the Effects of RAD1901 in the Treatment of Vasomotor Symptoms in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAD1901-002
Record Dates: First submitted 2009-03-06; First posted 2009-04-03 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Hot Flashes
Keywords: hot flashes; hot flushes; vasomotor symptoms; postmenopausal
MeSH Terms: conditions — Hot Flashes | interventions — RAD1901

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- RAD1901 10 mg (Experimental): Oral once a day for 28 days
  Interventions: Drug: RAD1901
- RAD1901 25 mg (Experimental): Oral once a day for 28 days
  Interventions: Drug: RAD1901
- RAD1901 50 mg (Experimental): Oral once a day for 28 days
  Interventions: Drug: RAD1901
- RAD1901 100 mg (Experimental): Oral once a day for 28 days
  Interventions: Drug: RAD1901
- Placebo (Placebo Comparator): Oral once a day for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAD1901 — 10 mg Oral once a day for 28 days.
  Arms: RAD1901 10 mg
Drug: RAD1901 — 25 mg Oral once a day for 28 days
  Arms: RAD1901 25 mg
Drug: RAD1901 — 50 mg Oral once a day for 28 days.
  Arms: RAD1901 50 mg
Drug: RAD1901 — 100 mg Oral once a day for 28 days
  Arms: RAD1901 100 mg
Drug: Placebo — Placebo Oral once a day for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether RAD1901 is effective in decreasing hot flashes in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Have documented evidence of a minimum of 7 moderate to severe hot flashes per day, or 50 per week.
2. Be in good general health as determined by medical history, physical examination, and inclusion procedures and is without evidence of any clinically significant abnormalities.
3. Have a normal pelvic assessment with no clinically significant signs on examination and pelvic ultrasound.
4. Have a normal mammogram at the time of study screening.

Exclusion Criteria:

1. A history of chronic or recurrent renal, hepatic, pulmonary, allergic, cardiovascular, gastrointestinal, endocrine, central nervous system, hematologic, immunologic or metabolic diseases to a degree that would compromise patient safety or interfere with the interpretation of study data. A history of active presence of thrombophlebitis, thrombosis, thromboembolic disorders.
2. A history of active presence of stroke, transient ischemic attack (TIA), heart attack or ischemic heart disease.
3. Unexplained vaginal bleeding within the 3 months prior to study entry.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Radius Health, Inc.
Locations (1):
- Radius Health, Inc., Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Hattersley G, Harris AG, Simon JA, Constantine GD. Clinical investigation of RAD1901, a novel estrogen receptor ligand, for the treatment of postmenopausal vasomotor symptoms: a phase 2 randomized, placebo-controlled, double-blind, dose-ranging, proof-of-concept trial. Menopause. 2017 Jan;24(1):92-99. doi: 10.1097/GME.0000000000000726. PMID 27575546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RAD1901 10 mg | RAD1901 25 mg | RAD1901 50 mg | RAD1901 100 mg | Placebo
Started | 22 | 20 | 21 | 18 | 19
Completed | 20 | 18 | 18 | 16 | 17
Not Completed | 2 | 2 | 3 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Inability to complete study procedures | 1 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Personal reason | 0 | 0 | 0 | 0 | 1
Not completed — Prohibited medication | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor decision | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAD1901 10 mg | RAD1901 25 mg | RAD1901 50 mg | RAD1901 100 mg | Placebo | Total
Number analyzed (Participants) | 22 | 20 | 21 | 18 | 19 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (5.74) | 55.2 (7.74) | 53.7 (5.68) | 55.7 (6.45) | 53.8 (5.74) | 54.3 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 21 | 18 | 19 | 100
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 22 | 20 | 21 | 18 | 19 | 100
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Frequency of Hot Flashes Over Time
Description: Percent change of moderate and severe hot flash frequency at 4 weeks compared to baseline using weekly Subject diary data, in the intent-to-treat population.
Time Frame: Week 4 minus baseline week
Population: The intent-to-treat population is defined as all patients who received one or more doses of study drug.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | RAD1901 10 mg | RAD1901 25 mg | RAD1901 50 mg | RAD1901 100 mg | Placebo
Number analyzed (Participants) | 22 | 20 | 21 | 18 | 19
Percent change from baseline | -77.2 (20.43) | -51.8 (45.02) | -53.8 (39.16) | -67.0 (33.85) | -54.1 (37.72)

2. Secondary Outcome: Determine the Effects of RAD1901 on Follicular Stimulating Hormone (FSH) Over Time.
Description: Percent change in FSH at Day 29 compared to baseline, in the intent-to-treat population.
Time Frame: Day 29 minus baseline
Population: The intent-to-treat (ITT) population is defined as all patients who received one or more doses of study drug. Based on patients who had a result on Day 29.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | RAD1901 10 mg | RAD1901 25 mg | RAD1901 50 mg | RAD1901 100 mg | Placebo
Number analyzed (Participants) | 20 | 18 | 18 | 16 | 17
Percent change from baseline | 4.24 (34.077) | -6.56 (13.933) | -4.42 (24.381) | -3.26 (11.373) | 8.67 (62.175)

3. Secondary Outcome: Determine the Effects of RAD1901 on Luteinizing Hormone (LH) Over Time.
Description: Percent change in LH levels at Day 29 compared to baseline, in the intent-to-treat population.
Time Frame: Day 29 minus baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | RAD1901 10 mg | RAD1901 25 mg | RAD1901 50 mg | RAD1901 100 mg | Placebo
Number analyzed (Participants) | 20 | 18 | 18 | 16 | 17
Percent change from baseline | -12.81 (27.551) | -0.19 (19.573) | -10.94 (22.609) | 3.57 (22.392) | 6.70 (36.270)

4. Primary Outcome: Percent Change in Composite Score Over Time
Description: Percent change in composite score (frequency x severity) of hot flashes (Mild=1, Moderate=2, Severe=3) at 4 weeks compared to baseline, in the intent-to-treat population.
Time Frame: Week 4 minus baseline week
Population: The intent-to-treat population is defined as all patients who received one or more doses of study drug.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | RAD1901 10 mg | RAD1901 25 mg | RAD1901 50 mg | RAD1901 100 mg | Placebo
Number analyzed (Participants) | 22 | 20 | 21 | 18 | 19
Percent change from baseline | -75.65 (18.655) | -55.48 (39.442) | -48.78 (39.806) | -66.21 (33.226) | -55.80 (35.523)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 2 months during this study; from start of treatment to the end-of-treatment visit (Day 29) and 30 days after end-of-treatment visit.
Description: Method of routinely determining whether or not certain adverse events have occurred was by regular investigator assessment and regular laboratory testing.
Arm/Group | RAD1901 10 mg | RAD1901 25 mg | RAD1901 50 mg | RAD1901 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/21 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 16/22 | 14/20 | 14/21 | 14/18 | 11/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD1901 10 mg (N=22) | RAD1901 25 mg (N=20) | RAD1901 50 mg (N=21) | RAD1901 100 mg (N=18) | Placebo (N=19)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Gastritis (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Salivary Gland Enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 4 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 1 | 0 | 1
Blood Triglyerides Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hypocholesterolaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Sensation of Heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Cluster Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 2 | 2 | 2 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Trigeminal Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Varicose Vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results may not be published prior to Study Report completion. Subsequent to formation of a Publications Committee, Investigators may publish results, providing a manuscript to Sponsor =/> 30 days prior to its submission. Sponsor will provide manuscript to Investigators =/> 30 days prior to its submission. Investigator will comply with Sponsor's policy, withholding publication for another 60 days to permit Sponsor to obtain patent or other proprietary rights protection, if deemed necessary.